CLINICAL TRIAL: NCT02280200
Title: Efficacy of Ankle-Foot Orthoses on Walking Ability in Peripheral Artery Disease: The AFO for PAD Trial I
Brief Title: Ankle-foot Orthoses for Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mays-2; U54GM104944 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Artery Disease
Keywords: claudication; ankle foot orthoses; community walking exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFO to improve outcomes (Experimental): Patients completed graded treadmill testing, followed by 12 weeks of unstructured community-based walking using the AFO ad libitum
  Interventions: Device: AFO to improve outcomes
- Historical Controls (No Intervention): Historical PAD control group (n = 10) received upfront advice to walk at home with no intervention

INTERVENTIONS:
Device: AFO to improve outcomes — Ankle foot orthoses (AFO) are light-weight, low profile carbon fiber devices that store and release energy during ambulation. The AFO, in combination with standard of care advice to walk more, will be used to determine if there is any improvement in PAD patient outcomes.
  Arms: AFO to improve outcomes

SUMMARY:
The primary aim of this study is to investigate the effect of an ankle foot orthoses (AFO) on the primary outcome of peak walking time (PWT) in patients with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The investigators will test the hypothesis that PAD patients using an AFO during a graded exercise test will demonstrate a greater PWT compared to PWT assessed without the use of an AFO. Secondary hypotheses include evaluation of the effect of an AFO on: 1) calf muscle function, 2) claudication onset time, 3) functional ability, 4) peak oxygen consumption, and 5) patient-reported outcomes. We will also examine the effects of the AFO on outcomes following 12 weeks of community walking.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with atherosclerotic peripheral arterial disease (PAD).
* Patients who experience calf claudication
* ≥40 years of age
* An abnormal ankle-brachial index (ABI) of ≤.90.
* For patients with an ABI >.90 and <1.00, a post-exercise ABI drop of 15% or more compared to the resting ABI

Exclusion Criteria:

* Lower extremity amputation(s) which interfere(s) with walking.
* Critical limb ischemia (i.e., ischemic rest pain, ulcers/gangrene on the lower extremities).
* Non-atherosclerotic PAD (e.g., popliteal entrapment syndrome, Takayasu's arteritis)
* Major surgical procedures that are contraindicated to an exercise program (e.g., recent organ transplant) or coronary artery bypass graft within 6 months prior to screening.
* Primarily limitations to exercise due to chronic obstructive pulmonary disease, angina or heart failure.
* Myocardial infarction within 3 months prior to screening.
* Acute coronary syndrome symptoms diagnosed at time of screening.
* Significant ischemic changes (documented on the 12-lead electrocardiogram) with horizontal or down-sloping ST-segment depression ≥ 0.5mm at rest and >1 mm with exercise in 3 beats for 2 contiguous leads, relative to the PR-segment (or ST-segment elevation ≥1mm).
* Transient ischemic attack or stroke 3 months prior to screening.
* New left bundle branch block or sustained ventricular tachycardia >30 seconds during screening.
* Uncontrolled hypertension defined as ≥180 systolic or ≥100 diastolic resting blood pressure during screening.
* Women who are pregnant (women of childbearing potential, a pregnancy test will be performed at screening.
* Individuals currently incarcerated.
* Evidence of acute impairment from alcohol or other illicit drugs.
* Lack of diabetes control (glycated hemoglobin >12%)
* Patients who are anemic (Hgb <11 g/dL for women and <10 g/dL for men).
* Any other clinically significant diseases (e.g., pulmonary, renal, psychiatric, immunological) that are not stabilized or may otherwise confound the results of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J. Mays, PhD, MPH, MS, Principal Investigator — International Heart Institute of Montana Foundation
Locations (1):
- International Heart Institute of Montana Foundation, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mays RJ, Mays AA, Mizner RL. Efficacy of ankle-foot orthoses on walking ability in peripheral artery disease. Vasc Med. 2019 Aug;24(4):324-331. doi: 10.1177/1358863X19831765. Epub 2019 Mar 29. PMID 30924412
- See also: Click here for more information about the sponsor — http://ctrin.unlv.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AFO to Improve Outcomes | Historical Controls
Started | 15 | 13
Completed | 12 | 10
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- AFO to Improve Outcomes: open label, non-interventional design (all patients who volunteer for trial receive AFO)
  AFO to improve outcomes: Ankle foot orthoses (AFO) are light-weight, low profile carbon fiber devices that store and release energy during ambulation. The AFO, in combination with standard of care advice to walk more, will be used to determine if there is any improvement in PAD patient outcomes.
- Total: Total of all reporting groups
Arm/Group | AFO to Improve Outcomes | Historical Controls | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (12.4) | 63.1 (6.7) | 65.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 14 | 5 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in WIQ Distance Subscore
Description: In the Walking Impairment Questionnaire distance subcategory, participants are asked to rate the degree of difficulty walking specific distances on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scale units
Arm/Group | AFO to Improve Outcomes | Historical Controls
Number analyzed (Participants) | 15 | 10
Scale units | 22.7 (24.5) | -7.2 (13.2)

2. Primary Outcome: Change in WIQ Speed Subscore
Description: In the Walking Impairment Questionnaire speed subcategory, participants are asked to rate the degree of difficulty walking one block at specific speeds, ranging from walking slowly to jogging, on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scale units
Arm/Group | AFO to Improve Outcomes | Historical Controls
Number analyzed (Participants) | 15 | 10
Scale units | 14.9 (17.1) | -7.5 (19.6)

3. Primary Outcome: Change in WIQ Stair-Climbing Subscore
Description: In the Walking Impairment Questionnaire stair-climbing subcategory, participants are asked to rate the degree of difficulty climbing a specified number of stair flights, ranging from 1 to 3 stair flights, on a graded scale of 0 to 4. A score of 0 indicates the inability to climb the flights specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent of score
Arm/Group | AFO to Improve Outcomes | Historical Controls
Number analyzed (Participants) | 15 | 10
percent of score | 18.9 (23.5) | 0 (37.2)

4. Primary Outcome: Change in SF-36 PCS
Description: Change in Medical Outcomes Study Short Form 36-item questionnaire, Physical Component Summary The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scale units
Arm/Group | AFO to Improve Outcomes | Historical Controls
Number analyzed (Participants) | 15 | 10
Scale units | 2.9 (5) | 2.1 (6.7)

5. Primary Outcome: Change in SF-36 MCS
Description: Change in Medical Outcomes Study Short Form 36-item questionnaire, Mental Component Summary The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scale units
Arm/Group | AFO to Improve Outcomes | Historical Controls
Number analyzed (Participants) | 15 | 10
Scale units | 4.3 (7.6) | -1.1 (6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | AFO to Improve Outcomes | Historical Controls
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/15 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AFO to Improve Outcomes (N=15) | Historical Controls (N=10)
Chronic Respiratory Problems (Respiratory, thoracic and mediastinal disorders) | 1 | 0
End-stage COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower Limb Skin Infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT02280200/Prot_SAP_000.pdf